CLINICAL TRIAL: NCT03368235
Title: A Phase 2a, Randomised, Double-blind, Parallel Study to Assess the Efficacy, Safety and Tolerability of AZD9567 Compared to Prednisolone 20 mg in Patients With Active Rheumatoid Arthritis (RA)
Brief Title: Early Phase Study to Assess Efficacy and Safety of AZD9567 Versus Prednisolone in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D6470C00003
Record Dates: First submitted 2017-11-03; First posted 2017-12-11 (Actual); Results first posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-08

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis, swollen joints, tender joints, autoimmunity
MeSH Terms: conditions — Arthritis, Rheumatoid; Autoimmune Diseases | interventions — AZD9567; Prednisolone

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, parallell arm study with two weeks treatment of AZD9567 or prednisolone
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double dummy technique
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZD9567 (Experimental): oral suspension of 40 mg AZD9567 once daily (OD) for two weeks
  Interventions: Drug: AZD9567
- Prednisolone (Active Comparator): oral OD treatment of 20 mg prednisolone administered as capsules
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: AZD9567 — oral OD SGRM administered as suspension
  Arms: AZD9567
Drug: Prednisolone — oral capsules of 20 mg prednisolone administered OD for two weeks
  Arms: Prednisolone

SUMMARY:
This is a phase 2a study to be run in 2-3 countries in European Union involving 5-6 sites. It will enroll approximately 80 patients to ensure 40 randomized with active rheumatoid arthritis. The treatment period is 2 weeks and total study duration per patient is approximately 1 month. The study drugs are AZD9567 40 mg (an oral SGRM) and the comparator is prednisolone 20mg. The primary endpoint is DAS28 including evaluation of 28 joints and C-reactive protein. Safety parameters will also be evaluated and a biomarker program is included for future research.

DETAILED DESCRIPTION:
This randomized double blind with double dummy technique phase 2a study will be run in 2-3 EU countries, most likely Sweden, Denmark and The Netherlands involving 5-6 sites. It is estimated that 80-100 patients have to be enrolled to ensure the randomization target of 40. The study population is patients with rheumatoid arthritis on stable treatment with conventional disease-modifying anti-rheumatic drugs (DMARDs) with an active flare. It is a two-arm parallel study and the randomization ratio is 1:1 to the two weeks of once daily treatment of 40 mg of AZD9567 and 20 mg prednisolone.

The primary objective is to assess the efficacy of AZD9567 40 mg, compared to prednisolone 20 mg in patients with active rheumatoid arthritis in spite of stable treatment with conventional and/or s.c/i.v. biological DMARDs and the primary variable is change from baseline in 28 joint Disease Activity Score using CRP (DAS28 - CRP). As secondary variables swollen and tenderness of 66-68 joints and safety variables are also included. For exploratively purposes there is also a biomarker program, collecting blood samples for future research.

ELIGIBILITY:
Inclusion Criteria:

1. Established RA diagnosis according to the 2010 American College of Rheumatology (ACR)/EULAR classification or the 1987 criteria
2. Active RA (DAS28-CRP score ≥ 3.2) with at least 3 swollen joints and 3 tender joints using the DAS28 joint count
3. Patients must have be on stable dosing of conventional and/or s.c./i.v biological DMARDs for the last 8 weeks prior to Visit 1
4. CRP levels >5mg/L at screening if seronegative for Rheumatoid Factor (RF) and Anti-Cyclic Citrullinated Peptide antibody (anti-CCP Ab), or >2mg/L if seropositive for either marker
5. BMI between 18 and 35 (inclusive)
6. Negative pregnancy test (serum) for female subjects of childbearing potential

Exclusion Criteria:

1. History or current inflammatory rheumatic disease other than RA (secondary Sjogren's syndrome excluded)
2. History or current clinically important disease which may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
3. Any clinical contraindications to treatment with steroids
4. Oral or parenteral steroids (beyond study medication) 8 weeks prior to study start and during the study. Stable use and dose of topical and inhaled steroids for longer than 4 w prior to randomization is acceptable
5. Use of any prohibited medication during the study or if the required washout time of such medication was not adhered to
6. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity to drugs with a similar class to study drugs
7. Any concomitant medications that are known to be associated with Torsades de Pointes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob M Van Laar, Professor, Principal Investigator — UMC Utrecht
Locations (5):
- Netherlands (3):
  - Research Site, Enschede
  - Research Site, Maastricht
  - Research Site, Utrecht
- Sweden (2):
  - Research Site, Gothenburg
  - Research Site, Lund

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Redacted Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6470C00003&attachmentIdentifier=935d5c96-53f7-4250-97cb-b99df948ee2e&fileName=D6470C00003_Protocol_v3.0_Redacted_19-03-2019.pdf&versionIdentifier=
- See also: SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6470C00003&attachmentIdentifier=271824b2-bcd4-4988-ae51-dbad237ee5d5&fileName=D6470C00003_Statistical_Analysis_Plan_28-11-2019.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 2a study conducted in participants with active rheumatoid arthritis (RA) in spite of stable treatment with conventional disease-modifying anti-rheumatic drugs at 5 investigational sites across Sweden and The Netherlands between 18 January 2018 and 12 November 2019.
Pre-assignment Details: A total of 21 participants were randomized in a 1:1 ratio to take either AZD9567 or prednisolone in a 2-week double-blind, double-dummy treatment period.
Groups:
- AZD9567: Participants received AZD9567 40 milligram (mg) oral suspension and placebo capsules matching with prednisolone, orally once daily, for 2 weeks.
- Prednisolone: Participants received prednisolone 20 mg oral capsules and placebo oral suspension matching with AZD9567, once daily for 2 weeks.
Period: Overall Study
Arm/Group | AZD9567 | Prednisolone
Started | 11 | 10
Completed | 11 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full analysis set (FAS) included all participants who were randomized and received at least 1 dose of study treatment.
Groups:
- AZD9567: Participants received AZD9567 40 mg oral suspension and placebo capsules matching with prednisolone, orally once daily, for 2 weeks.
- Total: Total of all reporting groups
Arm/Group | AZD9567 | Prednisolone | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (8.41) | 55.5 (13.58) | 60.2 (11.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Least Square (LS) Mean Change From Baseline in 28 Joint Disease Activity Score Using C-Reactive Protein (DAS28-CRP) at Day 15
Description: The DAS28-CRP is a measure of disease activity in RA. The score includes the number of tender and swollen joints (out of 28), CRP level (a measure of inflammation in the blood), and the patient's global assessment (PGA) of health (ranging from very well to very poor). The DAS28-CRP was derived as follows: 0.56 x √[tender joint count 28 (TJC28)] + 0.28 x √[swollen joint count 28 (SJC28)] + 0.014 x global health (GH) + 0.36 x Ln(CRP+1) + 0.96 to produce the overall DAS28-CRP score on a scale ranged from 0-10 with higher score indicating worse RA symptoms. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) prior to the first dose of study treatment.
Time Frame: Baseline (Day 1) and Day 15
Population: The FAS included all participants who were randomized and received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AZD9567 | Prednisolone
Number analyzed (Participants) | 11 | 10
score on a scale | -1.931 (0.3460) | -2.403 (0.3373)
Statistical Analysis 1: Comparison: AZD9567 vs Prednisolone; MMRM = mixed model repeated measures; Test type: Other; p = 0.315, MMRM — Based on MMRM model with the baseline DAS28-CRP score as a continuous covariate and country, visit and treatment group as categorical fixed effects, as well as visit interaction with treatment group, using unstructured covariance matrix; LS mean difference = 0.472, 95% CI 2-sided [-0.487 to 1.431], Standard Error of Mean 0.4569

2. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) 20, ACR50 and ACR70 Responses
Description: The ACR20, ACR50 or ACR70 was achieved if there was at least a 20%, 50% or 70% improvement from baseline in swollen joint count 66 (SJC66) and tender joint count 68 (TJC68) and 3 or more of the 5 following assessments: participant's assessment of pain, GH, physician's global assessment of disease activity, participant's assessment of physical function and CRP. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) prior to the first dose of study treatment.
Time Frame: Day 15
Population: The FAS included all participants who were randomized and received at least 1 dose of study treatment. Participants with missing ACR assessment at Day 15 were considered as non-responders in the respective analysis.
Measure: Number; unit: percentage of participants
Arm/Group | AZD9567 | Prednisolone
Number analyzed (Participants) | 11 | 10
percentage of participants
  ACR20 | 63.6 | 70.0
  ACR50 | 36.4 | 70.0
  ACR70 | 18.2 | 50.0
Statistical Analysis 1: Comparison: AZD9567 vs Prednisolone; Treatment comparison ACR20: AZD9567 Vs prednisolone; Test type: Other; p = 0.807, Regression, Logistic — Logistic regression model with the treatment group, country and baseline DAS28-CRP as covariate; Odds Ratio (OR) = 0.807, 95% CI 2-sided [0.12 to 5.34]
Statistical Analysis 2: Comparison: AZD9567 vs Prednisolone; Treatment comparison ACR50: AZD9567 Vs prednisolone; Test type: Other; p = 0.198, Fisher Exact
Statistical Analysis 3: Comparison: AZD9567 vs Prednisolone; Treatment comparison ACR70: AZD9567 Vs prednisolone; Test type: Other; p = 0.183, Fisher Exact

3. Secondary Outcome: LS Mean Change From Baseline in SJC66 Score at Day 15
Description: A total of 66 joints (33 left, 33 right) were evaluated for swelling. The swollen joint count represents the number of joints in which there was synovial fluid and or soft tissue swelling, but not if bony overgrowth was found. A swollen joint was scored as 0 (absent) and 1 (present) for each joint. The SJC66 was calculated as sum of swollen joints with present status on electronic case report form (eCRF). The swollen joint count ranged from 0-66 with higher score indicating disease severity. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) prior to the first dose of study treatment.
Time Frame: Baseline and Day 15
Population: The FAS included all participants who were randomized and received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AZD9567 | Prednisolone
Number analyzed (Participants) | 11 | 10
score on a scale | -6.24 (0.894) | -6.66 (0.860)
Statistical Analysis 1: Comparison: AZD9567 vs Prednisolone; Test type: Other; p = 0.717, MMRM — The MMRM with the baseline SJC66 score as a continuous covariate and country, visit and treatment group as categorical fixed effects, as well as visit interaction with treatment group, using unstructured covariance matrix; LS mean difference = 0.42, 95% CI 2-sided [-1.98 to 2.81], Standard Error of Mean 1.136

4. Secondary Outcome: LS Mean Change From Baseline in TJC68 Score at Day 15
Description: A total of 68 joints (34 left, 34 right) were evaluated for tenderness. The tender joint count represents the number of joints in which pain was reported. A tender joint was scored as 0 (absent) and 1 (present) for each joint. The TJC68 was calculated as sum of tender joints with present status on eCRF. The tender joint count ranged from 0-68 with higher score indicating disease severity. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) prior to the first dose of study treatment.
Time Frame: Baseline and Day 15
Population: The FAS included all participants who were randomized and received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AZD9567 | Prednisolone
Number analyzed (Participants) | 11 | 10
score on a scale | -9.02 (2.463) | -7.90 (2.362)
Statistical Analysis 1: Comparison: AZD9567 vs Prednisolone; Test type: Other; p = 0.724, MMRM — The MMRM with the baseline TJC68 score as a continuous covariate and country, visit and treatment group as categorical fixed effects, as well as visit interaction with treatment group, using unstructured covariance matrix; LS mean difference = -1.12, 95% CI 2-sided [-7.69 to 5.46], Standard Error of Mean 3.115

5. Secondary Outcome: LS Mean Change From Baseline in TJC28 Score at Day 15
Description: TJC28 was evaluated as one of the components that comprised the DAS28-score. A total of 28 joints (14 left, 14 right) were evaluated for tenderness as obtained from the joint count right or left eCRF. The tender joint count represents the number of joints in which pain was reported. A tender joint was scored as 0 (absent) and 1 (present) for each joint. The TJC28 was calculated as sum of tender joints with present status on eCRF. The tender joint count ranged from 0-28 with higher score indicating disease severity. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) prior to the first dose of study treatment.
Time Frame: Baseline and Day 15
Population: The FAS included all participants who were randomized and received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AZD9567 | Prednisolone
Number analyzed (Participants) | 11 | 10
score on a scale | -6.12 (1.251) | -6.07 (1.208)
Statistical Analysis 1: Comparison: AZD9567 vs Prednisolone; Test type: Other; p = 0.973, MMRM — The MMRM with the baseline TJC28 score as a continuous covariate and country, visit and treatment group as categorical fixed effects, as well as visit interaction with treatment group, using unstructured covariance matrix; LS mean difference = -0.05, 95% CI 2-sided [-3.43 to 3.32], Standard Error of Mean 1.600

6. Secondary Outcome: LS Mean Change From Baseline in SJC28 Score at Day 15
Description: SJC28 was evaluated as one of the components that comprised the DAS28-score. A total of 28 joints (14 left, 14 right) were evaluated for swelling as obtained from the joint count right or left eCRF. The swollen joint count represents the number of joints in which there was synovial fluid and or soft tissue swelling, but not if bony overgrowth was found. A swollen joint was scored as 0 (absent) and 1 (present) for each joint. The SJC28 was calculated as sum of swollen joints with present status on eCRF. The swollen joint count ranged from 0-28 with higher score indicating disease severity. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) prior to the first dose of study treatment.
Time Frame: Baseline and Day 15
Population: The FAS included all participants who were randomized and received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AZD9567 | Prednisolone
Number analyzed (Participants) | 11 | 10
score on a scale | -5.14 (0.653) | -5.40 (0.628)
Statistical Analysis 1: Comparison: AZD9567 vs Prednisolone; Test type: Other; p = 0.757, MMRM — The MMRM with the baseline SJC28 score as a continuous covariate and country, visit and treatment group as categorical fixed effects, as well as visit interaction with treatment group, using unstructured covariance matrix; LS mean difference = 0.26, 95% CI 2-sided [-1.50 to 2.03], Standard Error of Mean 0.837

7. Secondary Outcome: LS Mean Change From Baseline in GH Score at Day 15
Description: GH was evaluated as one of the components that comprised the DAS28-score. Participant's GH was measured using PGA of disease activity by means of the visual analogue scale (VAS). The PGA VAS consists of a 100 millimeter (mm) long scale ranging from 0 (very well) to 100 (very poor). Higher score indicated greater disease severity. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) prior to the first dose of study treatment.
Time Frame: Baseline and Day 15
Population: The FAS included all participants who were randomized and received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AZD9567 | Prednisolone
Number analyzed (Participants) | 11 | 10
score on a scale | -27.7 (7.26) | -37.4 (7.11)
Statistical Analysis 1: Comparison: AZD9567 vs Prednisolone; Test type: Other; p = 0.325, MMRM — The MMRM with the baseline GH score as a continuous covariate and country, visit and treatment group as categorical fixed effects, as well as visit interaction with treatment group, using unstructured covariance matrix; LS mean difference = 9.8, 95% CI 2-sided [-10.5 to 30.1], Standard Error of Mean 9.67

8. Secondary Outcome: LS Mean Change From Baseline in CRP at Day 15
Description: CRP was evaluated as one of the components that comprised the DAS28-score. The CRP was collected at the local laboratory during screening and central laboratory on Days 1, 8, 15 and 28. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) prior to the first dose of study treatment.
Time Frame: Baseline and Day 15
Population: The FAS included all participants who were randomized and received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: mg per liter (L)
Arm/Group | AZD9567 | Prednisolone
Number analyzed (Participants) | 11 | 10
mg per liter (L) | -10.830 (2.4207) | -15.586 (2.5245)
Statistical Analysis 1: Comparison: AZD9567 vs Prednisolone; Test type: Other; p = 0.187, MMRM — The MMRM with the baseline CRP score as a continuous covariate and country, visit and treatment group as categorical fixed effects, as well as visit interaction with treatment group, using unstructured covariance matrix; LS mean difference = 4.756, 95% CI 2-sided [-2.514 to 12.025], Standard Error of Mean 3.4725

9. Secondary Outcome: LS Mean Change From Baseline in Participant's Assessment of Pain Score at Day 15
Description: Participant's assessment of pain score was evaluated as one of the components that comprised the ACR. Participant's assessment of pain score was assessed from the amount of pain due to RA on a VAS ranging from 0 (no pain) to 100 (extreme pain). Higher score indicated greater disease severity. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) prior to the first dose of study treatment.
Time Frame: Baseline and Day 15
Population: The FAS included all participants who were randomized and received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AZD9567 | Prednisolone
Number analyzed (Participants) | 11 | 10
score on a scale | -27.3 (8.17) | -43.4 (7.71)
Statistical Analysis 1: Comparison: AZD9567 vs Prednisolone; Test type: Other; p = 0.144, MMRM — The MMRM with the baseline participant's assessment of pain score as a continuous covariate and country, visit and treatment group as categorical fixed effects, as well as visit interaction with treatment group, using unstructured covariance matrix; LS mean difference = 16.0, 95% CI 2-sided [-6.0 to 38.1], Standard Error of Mean 10.49

10. Secondary Outcome: LS Mean Change From Baseline in Physician's Global Assessment of Disease Activity Score at Day 15
Description: Physician's global assessment of disease activity score was evaluated as one of the components that comprised the ACR. The physician's global assessment of disease activity was measured on a VAS ranging from 0 (very well) to 100 (very poor). Higher score indicated greater disease severity. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) prior to the first dose of study treatment.
Time Frame: Baseline and Day 15
Population: The FAS included all participants who were randomized and received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AZD9567 | Prednisolone
Number analyzed (Participants) | 11 | 10
score on a scale | -37.0 (4.38) | -40.9 (4.30)
Statistical Analysis 1: Comparison: AZD9567 vs Prednisolone; Test type: Other; p = 0.512, MMRM — The MMRM with the baseline disease activity score as a continuous covariate and country, visit and treatment group as categorical fixed effects, as well as visit interaction with treatment group, using unstructured covariance matrix; LS mean difference = 3.8, 95% CI 2-sided [-8.3 to 16.0], Standard Error of Mean 5.73

11. Secondary Outcome: LS Mean Change From Baseline in Participant's Assessment of Physical Function Score at Day 15
Description: Participant's assessment of physical function score was evaluated as one of the components that comprised the ACR. The participant's assessment of physical function across 8 functional areas was measured by health assessment questionnaire. The total score ranging from 0 (no difficulty) to 24 (inability to perform tasks). Higher score indicated greater disease severity. Baseline was defined as the last non-missing assessment (scheduled or unscheduled) prior to the first dose of study treatment.
Time Frame: Baseline and Day 15
Population: The FAS included all participants who were randomized and received at least 1 dose of study treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AZD9567 | Prednisolone
Number analyzed (Participants) | 11 | 10
score on a scale | -0.441 (0.1758) | -0.571 (0.1712)
Statistical Analysis 1: Comparison: AZD9567 vs Prednisolone; Test type: Other; p = 0.589, MMRM — The MMRM with the baseline physical function score as a continuous covariate and country, visit and treatment group as categorical fixed effects, as well as visit interaction with treatment group, using unstructured covariance matrix; LS mean difference = 0.131, 95% CI 2-sided [-0.370 to 0.631], Standard Error of Mean 0.2381

12. Secondary Outcome: Area Under the Plasma Concentration-Time Curve Until the Last Quantifiable Concentration (AUClast) of AZD9567
Description: The AUClast was determined using non-compartmental method and calculated using the linear trapezoidal rule when concentrations were increased and the logarithmic trapezoidal rule when concentrations were decreased.
Time Frame: Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4 and 6 hour postdose on Day 15.
Population: The Pharmacokinetic (PK) analysis set included all participants with at least 1 quantifiable AZD9567 concentration with a documented related dosing history.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanomole per L (h*nmol/L)
Arm/Group | AZD9567
Number analyzed (Participants) | 11
hour*nanomole per L (h*nmol/L) | 17800 (35.02)

13. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to 6 Hours After Dose (AUC0-6) of AZD9567
Description: The AUC0-6 was determined using non-compartmental method and calculated using the linear trapezoidal rule when concentrations were increased and the logarithmic trapezoidal rule when concentrations were decreased.
Time Frame: Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4 and 6 hour postdose on Day 15.
Population: The PK analysis set included all participants with at least 1 quantifiable AZD9567 concentration with a documented related dosing history.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*nmol/L
Arm/Group | AZD9567
Number analyzed (Participants) | 11
h*nmol/L | 17740 (35.34)

14. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of AZD9567
Description: The Cmax of AZD9567 was determined using non-compartmental method.
Time Frame: Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4 and 6 hour postdose on Day 15.
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | AZD9567
Number analyzed (Participants) | 11
nmol/L | 4468 (26.89)

15. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of AZD9567
Description: The tmax of AZD9567 was determined using non-compartmental method.
Time Frame: Predose and 0.25, 0.5, 1, 1.5, 2, 3, 4 and 6 hour postdose on Day 15.
Population: as for outcome 13
Measure: Median (Full Range); unit: hour
Arm/Group | AZD9567
Number analyzed (Participants) | 11
hour | 0.67 [0.33 to 1.03]

16. Secondary Outcome: Last Plasma Concentration Measured Before the Last Dose (Ctrough) of AZD9567
Description: The Ctrough of AZD9567 was determined using non-compartmental method before the last dose on Day 15.
Time Frame: Predose on Day 15
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | AZD9567
Number analyzed (Participants) | 11
nmol/L | NA (95.67) — Not calculable due to a zero predose value.

ADVERSE EVENTS:
Time Frame: From first administration of study treatment (Day 1) up to 2 weeks after last administration of study treatment, approximately 28 days.
Description: The Safety analysis set included all participants who were randomized and received at least 1 dose of study treatment.
Arm/Group | AZD9567 | Prednisolone
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/10
Other Adverse Events (participants affected / at risk) | 10/11 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9567 (N=11) | Prednisolone (N=10)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9567 (N=11) | Prednisolone (N=10)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 1 (2) | 0 (0)
Eye pain (Eye disorders) | 2 (3) | 0 (0)
Periorbital swelling (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Mood swings (Psychiatric disorders) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT03368235/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-28): https://cdn.clinicaltrials.gov/large-docs/35/NCT03368235/SAP_001.pdf